CLINICAL TRIAL: NCT04458259
Title: A PHASE 1, OPEN-LABEL, MULTI-CENTER, DOSE-FINDING, PHARMACOKINETIC, SAFETY AND TOLERABILITY STUDY OF PF 07265807 IN PARTICIPANTS WITH SELECTED ADVANCED OR METASTATIC SOLID TUMOR MALIGNANCIES
Brief Title: Study of PF-07265807 in Participants With Metastatic Solid Tumors.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Pfizer has made an internal business decision to not continue further development of PF-07265807. This decision was not due to major safety concerns or requests from any regulatory authorities.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C4201002; 2021-004270-59 (EudraCT Number); ARRAY-067-102 (Other: Alias Study Number)
Record Dates: First submitted 2020-06-24; First posted 2020-07-07 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Neoplasm Metastasis
Keywords: TAMK (TAM kinase); MER (mer proto-oncogene); MERTK (mer proto-oncogene tyrosine kinase); AXL (AXL receptor tyrosine kinase); AXL/MER; Selective kinase inhibitor; PD-1 (programmed cell death protein 1); PD-L1 (programmed cell death ligand 1); Immune modulator; Advanced Cancer; Metastatic Cancer; Solid Tumor Cancer; Metastatic Solid Tumor; Cervical Cancer; Gastric Cancer; Esophageal Cancer; Endometrial Cancer; Hepatocellular carcinoma (HCC); Melanoma; Merkel Cell Carcinoma; High levels of MicroSatellite Instability deficient MisMatch Repair (MSI-H-dMMR) tumor; Non-small cell lung cancer (NSCLC); Small cell lung cancer (SCLC); Renal cell carcinoma (RCC); Urothelial carcinoma; Colorectal cancer (CRC)
MeSH Terms: conditions — Neoplasm Metastasis; Parkinson Disease 4, Autosomal Dominant Lewy Body; Uterine Cervical Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Endometrial Neoplasms; Carcinoma, Hepatocellular; Melanoma; Carcinoma, Merkel Cell; Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Carcinoma, Renal Cell; Carcinoma, Transitional Cell; Colorectal Neoplasms | interventions — Axitinib

STUDY DESIGN:
Intervention Model Description: Dose escalation and expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Monotherapy Dose Escalation: Part 1 (Experimental): Monotherapy dose escalation of PF-07265807 in participants with select tumor types.
  Interventions: Drug: PF-07265807
- Doublet Dose Escalation: Part 2 (Experimental): Doublet combination dose escalation of PF-07265807 with sasanlimab in participants with select tumor types. PF-07265807 will dose escalate. Sasanlimab dose will stay constant.
  Interventions: Drug: PF-07265807; Drug: Sasanlimab
- Triplet Dose Escalation: Part 3 (Experimental): Triplet combination dose escalation of PF-07265807 with sasanlimab plus axitinib in participants with select tumor types. PF-07265807 will dose escalate. Sasanlimab dose will stay constant. Axitinib dose will follow label.
  Interventions: Drug: PF-07265807; Drug: Sasanlimab; Drug: Axitinib
- Expansion Phase: Part 4, Cohort 1 (Experimental): PF-07265807 monotherapy in participants with METex14 mutant NSCLC.
  Interventions: Drug: PF-07265807
- Expansion Phase: Part 4, Cohort 2 (Experimental): PF-07265807 with sasanlimab in participants with MSS CRC
  Interventions: Drug: PF-07265807; Drug: Sasanlimab
- Expansion Phase: Part 4, Cohort 3 (Experimental): PF-07265807 with sasanlimab in participants with PD-L1+ gastric cancer/GEJ
  Interventions: Drug: PF-07265807; Drug: Sasanlimab
- Expansion Phase: Part 4, Cohort 4 (Experimental): PF-07265807 with sasanlimab plus axitinib in participants with RCC
  Interventions: Drug: PF-07265807; Drug: Sasanlimab; Drug: Axitinib

INTERVENTIONS:
Drug: PF-07265807 — Given 2 weeks on/1 week off
  Other Names: ARRY-067
Drug: Sasanlimab — Given SC Q3W
  Other Names: PF-06801591; RN-888
  Arms: Doublet Dose Escalation: Part 2; Expansion Phase: Part 4, Cohort 2; Expansion Phase: Part 4, Cohort 3; Expansion Phase: Part 4, Cohort 4; Triplet Dose Escalation: Part 3
Drug: Axitinib — Dosed per package label starting with 5 mg PO BID
  Other Names: AG-013736; Inlyta
  Arms: Expansion Phase: Part 4, Cohort 4; Triplet Dose Escalation: Part 3

SUMMARY:
A First-in-Human Pharmacokinetic, Safety, and Tolerability Study of PF-07265807 as Monotherapy and in Combination in Participants with Advanced or Metastatic Solid Tumors

ELIGIBILITY:
Inclusion Criteria:

* At least one measurable (Parts 1-4) or non-measurable lesion (Parts 1-3), not previously irradiated, as defined by RECIST 1.1
* ECOG Performance Status 0 or 1, 2 with approval
* Adequate Bone Marrow Function
* Adequate Renal Function
* Adequate Liver Function
* Resolved acute effects of any prior therapy
* Able to provide adequate archival tumor tissue or freshly obtained tumor tissue (some participants will require mandatory pre- and on-treatment biopsy is part of the biomarker cohort).
* Life expectancy of at least 3 months.
* Part 1 and Part 2: Participants who are intolerant or resistant to standard treatment for selected solid tumors.
* Part 3: Participants with advanced/metastatic RCC with a clear cell component and progressed with no standard therapy available.
* Part 4, Cohort 1: Participants with NSCLC with METex14-skipping alteration(s) and progressed on at least 1 prior therapy.
* Part 4, Cohort 2: Participants with MSS CRC with intermediate TMB and progressed with no satisfactory alternative treatment available, but has not received prior treatment with an anti-PD-(L)1 therapy.
* Part 4, Cohort 3: Participants with metastatic gastric or GEJ adenocarcinoma that is PD-L1 positive that has progressed on at least 2 but no more than 3 prior chemotherapy regiments, but has not received prior treatment with an anti-PD-(L)1 therapy.
* Part 4, Cohort 4: Participants with metastatic RCC with a clear cell component with IMDC intermediate or poor risk that have not received any prior systemic therapy for metastatic disease.

Exclusion Criteria:

* Known active uncontrolled or symptomatic CNS metastases.
* Any other active malignancy within 2 years prior to enrollment.
* Major surgery within 6 weeks, radiation therapy within 4 weeks, systemic anti-cancer therapy within 2 week or 5 half-lives (4 weeks or 5 half-lives for antibody therapies or investigational drug(s) taken on another study) prior to study entry.
* Active or history of autoimmune disease requiring >10mg/day prednisone or other concurrent immunosuppressive therapy.
* Active, uncontrolled infection (controlled HBV, HCV, HIV/AIDS may be allowed) as defined in protocol.
* Retinal or other serious ophthalmic disorders as defined in protocol.
* Clinically significant cardiac disease as defined in protocol.
* Uncontrolled HTN that cannot be controlled by medications.
* Inability to consume or absorb study drug.
* Known or suspected hypersensitivity to PF-07265807.
* Prohibited concomitant medications as defined in protocol.
* Active inflammatory GI disease, uncontrollable chronic diarrhea, or previous gastric resection or lap band surgery affecting absorption.
* Active bleeding disorder.
* Discontinuation of prior checkpoint inhibitor for treatment-related toxicity.
* Experienced >= G3 treatment-related irAE with prior PD-(L)1 agent.
* Prior treatment with selective AXL/MERTK inhibitors

For participants receiving sasanlimab:

- Known history of non-infectious pneumonitis that required steroid treatment or current pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Parts 1, 2, and 3: Number of participants with dose limiting toxicities (DLTs) | Baseline through day 21 or 42
  DLTs will be evaluated during the first cycle (day 21) or two cycles (day 42). The number of DLTs will be used to determine the maximum tolerated dose (MTD)
Parts 1, 2 and 3: Number of participants with treatment emergent adverse events (AEs) | Baseline through approximately 2 years
  AEs as characterized by type, frequency, severity, timing, seriousness, and relationship to study therapy
Parts 1, 2, and 3: Number of participants with laboratory abnormalities | Baseline through approximately 2 years
  Laboratory abnormalities as characterized by type, frequency, severity, and timing.
Part 4: Overall Response Rate (ORR) | Baseline through approximately 2 years
  Response will be evaluable via radiographical tumor assessment by RECIST v1.1
Part 4, Cohort 4: Complete Response (CR) | Baseline through approximately 2 years
  Response will be evaluated via radiographical tumor assessment by RECIST v1.1

SECONDARY OUTCOMES:
Parts 1, 2, and 3: Maximum plasma concentration (Cmax) of PF-07265807 and its metabolite | Each cycle is 21 days. Cycle 1 Days 1 and 14, predose, 0.5,1,2,4,8 and 24 (if daily dosing) hours post dose; Cycle 1 Day 7, Cycle 2 Days 1 and 14 predose and 2 hours post dose; Cycle 3 Days 1 and 14 predose
  Single dose (Cmax) and multiple dose (assuming steady state is achieved; Cmax,ss) pharmacokinetic (PK) parameters of PF-07265807 and its metabolite
Parts 2 and 3: Maximum plasma concentration (Cmax) of sasanlimab | Through study completion, an average of 1 year
  Single dose (Cmax) pharmacokinetic (PK) parameters of sasanlimab
Part 3: Maximum plasma concentration at steady state (Cmax,ss) of axitinib | Each cycle is 21 days. Cycle 1 Day 1 predose; Cycle 1 Day 14 predose, 0.5,1,2,4, and 8 hours post dose
  Multiple dose (assuming steady state is achieved; Cmax,ss) pharmacokinetic (PK) parameters of axitinib
Parts 1, 2, and 3: Time to reach maximum plasma concentration (Tmax) of PF-07265807 and its metabolite | Each cycle is 21 days. Cycle 1 Days 1 and 14, predose, 0.5,1,2,4,8 and 24 (if daily dosing) hours post dose; Cycle 1 Day 7, Cycle 2 Days 1 and 14 predose and 2 hours post dose; Cycle 3 Days 1 and 14 predose
  Single dose (Tmax) and multiple dose (assuming steady state is achieved; Tmax,ss) pharmacokinetic parameters of PF-07265807 and its metabolite
Parts 2 and 3: Time to reach maximum plasma concentration (Tmax) of sasanlimab | Through study completion, an average of 1 year
  Single dose (Tmax) pharmacokinetic parameters of sasanlimab
Part 3: Time to reach maximum plasma concentration at steady state (Tmax,ss) of axitinib | Each cycle is 21 days. Cycle 1 Day 1 predose; Cycle 1 Day 14 predose, 0.5,1,2,4, and 8 hours post dose
  Multiple dose (assuming steady state is achieved; Tmax,ss) pharmacokinetic parameters of axitinib
Parts 1, 2, and 3: Area under the curve from the time of dose to the last measurable concentration (AUClast) of PF-07265807 and its metabolite | Each cycle is 21 days. Cycle 1 Days 1 and 14, predose, 0.5,1,2,4,8 and 24 (if daily dosing) hours post dose; Cycle 1 Day 7, Cycle 2 Days 1 and 14 predose and 2 hours post dose; Cycle 3 Days 1 and 14 predose
  Single dose (AUClast) pharmacokinetic parameters of PF-07265807 and its metabolite
Parts 2 and 3: Area under the curve from the time of dose to the last measurable concentration (AUClast) of sasanlimab | Through study completion, an average of 1 year
  Single dose (AUClast) pharmacokinetic parameters of sasanlimab
Parts 1, 2, and 3: Area under the curve from the time of dose to the time of the subsequent dose (AUCtau) at steady state of PF-07265807 and its metabolite | Each cycle is 21 days. Cycle 1 Days 1 and 14, predose, 0.5,1,2,4,8 and 24 (if daily dosing) hours post dose; Cycle 1 Day 7, Cycle 2 Days 1 and 14 predose and 2 hours post dose; Cycle 3 Days 1 and 14 predose
  Multiple dose assuming steady state is achieved (AUCtau,ss) pharmacokinetic parameters of PF-07265807 and its metabolite
Part 3: Area under the curve from the time of dose to the time of the subsequent dose (AUCtau) at steady state of axitinib | Each cycle is 21 days. Cycle 1 Day 1 predose; Cycle 1 Day 14 predose, 0.5,1,2,4, and 8 hours post dose
  Multiple dose assuming steady state is achieved (AUCtau,ss) pharmacokinetic parameters of axitinib
Parts 1, 2, and 3: Terminal elimination half-life (t1/2) of PF-07265807 and its metabolite | Each cycle is 21 days. Cycle 1 Days 1 and 14, predose, 0.5,1,2,4,8 and 24 (if daily dosing) hours post dose; Cycle 1 Day 7, Cycle 2 Days 1 and 14 predose and 2 hours post dose; Cycle 3 Days 1 and 14 predose
  As data permits, single dose (t1/2) pharmacokinetic parameters of PF-07265807 and its metabolite
Parts 2 and 3: Terminal elimination half-life (t1/2) of sasanlimab | Through study completion, an average of 1 year
  As data permits, single dose (t1/2) pharmacokinetic parameters of sasanlimab
Parts 1, 2, and 3: Area under the curve from the time of dose extrapolated to infinity (AUCinf) of PF-07265807 and its metabolite | Each cycle is 21 days. Cycle 1 Days 1 and 14, predose, 0.5,1,2,4,8 and 24 (if daily dosing) hours post dose; Cycle 1 Day 7, Cycle 2 Days 1 and 14 predose and 2 hours post dose; Cycle 3 Days 1 and 14 predose
  As data permits, single dose (AUCinf) pharmacokinetic parameters of PF-07265807 and its metabolite
Parts 2 and 3: Area under the curve from the time of dose extrapolated to infinity (AUCinf) of sasanlimab | Through study completion, an average of 1 year
  As data permits, single dose (AUCinf) pharmacokinetic parameters of sasanlimab
Parts 1, 2, and 3: Apparent oral clearance (CL/F) of PF-07265807 | Each cycle is 21 days. Cycle 1 Days 1 and 14, predose, 0.5,1,2,4,8 and 24 (if daily dosing) hours post dose; Cycle 1 Day 7, Cycle 2 Days 1 and 14 predose and 2 hours post dose; Cycle 3 Days 1 and 14 predose
  As data permits, single dose (CL/F) and multiple dose pharmacokinetic parameters of PF-07265807
Parts 2 and 3: Apparent clearance (CL/F) of sasanlimab | Through study completion, an average of 1 year
  As data permits, single dose (CL/F) pharmacokinetic parameters of sasanlimab
Parts 1, 2, and 3: Apparent terminal volume of distribution (Vz/F) of PF-07265807 | Each cycle is 21 days. Cycle 1 Days 1 and 14, predose, 0.5,1,2,4,8 and 24 (if daily dosing) hours post dose; Cycle 1 Day 7, Cycle 2 Days 1 and 14 predose and 2 hours post dose; Cycle 3 Days 1 and 14 predose
  As data permits, single dose (Vz/F) and multiple dose (Vss/F) pharmacokinetic parameters of PF-07265807
Parts 2 and 3: Apparent terminal volume of distribution (Vz/F) of sasanlimab | Through study completion, an average of 1 year
  As data permits, single dose (Vz/F) pharmacokinetic parameters of sasanlimab
Parts 1, 2, and 3: ORR | Baseline through approximately 2 years
  Response will be evaluable via radiographical tumor assessment by RECIST v1.1
Part 4: Number of participants with treatment emergent AEs | Baseline through approximately 2 years
  AEs as characterized by type, frequency, severity, timing, seriousness, and relationship to study therapy
Part 4: Number of participants with laboratory abnormalities | Baseline through approximately 2 years
  Laboratory abnormalities as characterized by type, frequency, severity, and timing
Part 4: Trough concentration (Ctrough) of PF-07265807 and its metabolite | Each cycle is 21 days. Cycle 1 Days 1 and 14 predose, 2, 4 hours post dose; Cycle 1 Day 7 predose and 2 hours post dose; Cycle 2 Days 1 and 14 predose
  Predose (Ctrough) pharmacokinetic (PK) parameter of PF-07265807 and its metabolite
Part 4: Post dose concentration (Cmax) of PF-07265807 and its metabolite | Each cycle is 21 days. Cycle 1 Days 1 and 14 predose, 2, 4 hours post dose; Cycle 1 Day 7 predose and 2 hours post dose; Cycle 2 Days 1 and 14 predose
  Post dose (Cmax) pharmacokinetic (PK) parameter of PF-07265807 and its metabolite
Part 4, Cohorts 2, 3 and 4: Trough concentration (Ctrough) of sasanlimab | Each cycle is 21 days. Cycle 1 Days 1, 7, and 14, Cycle 2 Day 1, Cycle 7 Day 1, and every 6 cycles thereafter predose
  Predose (Ctrough) pharmacokinetic (PK) parameter of sasanlimab
Part 4, Cohort 4: Trough concentration (Ctrough) of axitinib | Each cycle is 21 days. Cycle 1 Day 1 predose; Cycle 1 Day 14 predose, 2, and 4 hours post dose
  Predose (Ctrough) pharmacokinetic (PK) parameter of axitinib
Parts 2, 3, and 4 Cohorts 2-4: Immunogenicity of sasanlimab when given in combination | Through study completion, an average of 1 year
  Incidence and titer of anti-sasanlimab ADA response
Duration of Response | Baseline through approximately 2 years
  Response will be evaluable via radiographical tumor assessment by RECIST v1.1
Disease Control Rate | Baseline through approximately 2 years
  Response will be evaluable via radiographical tumor assessment by RECIST v1.1
Progression Free Survival | Baseline through approximately 2 years
  Response will be evaluable via radiographical tumor assessment by RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (30):
- United States (22):
  - Henry Eye Clinic, Fayetteville, Arkansas
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Highlands Oncology Group, Rogers, Arkansas
  - Highlands Oncology Group, Springdale, Arkansas
  - UCI Chao Family Comprehensive Cancer Center, Orange, California
  - Clinical & Translational Science Institute, San Francisco, California
  - UCSF Helen Diller Family Comprehensive Cancer Center - Mission Hall, San Francisco, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Rocky Mountain Lions Eye Institute (RMLEI), Aurora, Colorado
  - University of Colorado Hospital - Anschutz Cancer Pavilion (ACP), Aurora, Colorado
  - University of Colorado Hospital - Anschutz Inpatient Pavilion (AIP), Aurora, Colorado
  - University of Colorado Hospital - Anschutz Outpatient Pavilion (AOP), Aurora, Colorado
  - Community Health Network, Inc., Indianapolis, Indiana
  - Community Health Network Cancer Center North, Indianapolis, Indiana
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer Institute - Chestnut Hill, Newton, Massachusetts
  - Hackensack University Medical Center, Hackensack, New Jersey
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Duke Eye Center, Durham, North Carolina
  - Duke University Medical Center, lnvestigational Chemotherapy Service, Durham, North Carolina
  - The University of Texas M. D. Anderson Cancer Center, Houston, Texas
- University Health Network, Toronto, Ontario, Canada
- Italy (3):
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore, Roma, ROME
  - Istituto Nazionale Tumori IRCCS Fondazione Giovanni Pascale, Napoli
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore, Roma
- National Cancer Center Hospital East, Kashiwa, Chiba, Japan
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Fundacion Jimenez Díaz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4201002